CLINICAL TRIAL: NCT00131677
Title: Phase II Extended Safety Study of Tenofovir Disoproxil Fumarate (TDF) Among HIV-1 Negative Men
Brief Title: Extended Safety Study of Tenofovir Disoproxil Fumarate (TDF) Among HIV-1 Negative Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: San Francisco Department of Public Health (Other Government); AIDS Research Consortium of Atlanta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CDC-NCHHSTP-4323
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2013-08

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- active immediate (Active Comparator): participants in this arm start study product immediately upon enrollment
  Interventions: Drug: tenofovir disoproxil fumarate
- placebo immediate (Placebo Comparator): participants in this arm start study product immediately upon enrollment
  Interventions: Drug: placebo
- active delayed (Active Comparator): persons in this arm start study product 9 months after enrollment
  Interventions: Drug: tenofovir disoproxil fumarate
- placebo delayed (Placebo Comparator): participants in this arm start study product nine months after enrollment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tenofovir disoproxil fumarate — study product taken daily
  Other Names: Viread
  Arms: active delayed; active immediate
Drug: placebo — study product taken daily
  Arms: placebo delayed; placebo immediate

SUMMARY:
The purpose of this study is to examine safety and tolerability of daily tenofovir use in HIV-uninfected men.

DETAILED DESCRIPTION:
This study will assess the clinical and behavioral safety and tolerability of oral daily TDF use as pre-exposure prophylaxis (PrEP) to prevent HIV infection in uninfected men.

ELIGIBILITY:
Inclusion Criteria:

* Healthy biologic male (male at birth)
* 18-60 years of age
* HIV-1 negative by licensed, commercially available, FDA-approved whole blood rapid enzyme immunoassay (EIA) at screening and enrollment
* Reports any anal sex with a man in the last 12 months
* Able to understand and pass comprehension assessment questionnaire
* Able to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* Able to understand English
* Adequate renal function: calculated creatinine clearance of at least 70 mL/min
* Hepatic transaminases (AST and ALT) less than or equal to 2x upper limit of normal (ULN)
* Total bilirubin less than or equal to 1.5 mg/dL
* Absolute neutrophil count at least 1,500/mm3;
* Platelets at least 100,000/mm3;
* Hemoglobin at least 9.5 g/dL
* Serum amylase less than or equal to 1.5 x ULN
* Biochemical profile: within normal limits for serum phosphorus, potassium, sodium, and calcium.
* Hepatitis B surface antigen negative
* Normal urine dipstick or urinalysis (UA)

Exclusion Criteria:

* Active untreated syphilis
* Current uncontrolled hypertension (blood pressure > 160/100 mmHg)
* Mutually monogamous for > one year with a known HIV antibody negative partner
* History of chronic renal disease, known osteoporosis, osteomalacia, or osteopenia
* Current or expected participation in other longitudinal HIV behavioral or biomedical research study
* Current HIV antiretroviral use
* Receiving or planning to receive on-going therapy with any nephrotoxic agents or experimental/investigational agents
* Previous or expected requirements for the administration of immunosuppressive/ immunomodulatory therapy (e.g. chronic systemic steroids, interferon, interleukins, chemotherapy, radiation).
* Evidence of a gastrointestinal malabsorption syndrome or chronic nausea or vomiting which may confer an inability to receive an orally administered medication.
* Current alcohol or substance abuse judged by the investigator to potentially interfere with participant compliance.
* Imminently life-threatening medical conditions (malignancy, immunosuppressive disease [e.g. lymphoma]), or other serious disease or conditions (e.g. cardiovascular, renal, diabetes) within the last 5 years or that are unstable and/or require chronic medication that would impede compliance with study requirements and complicate the interpretation of adverse events
* Expected to be non-compliant with study visits or planning to move within 24 months to an area where the study will not be conducted
* Any other clinical or social condition, prior therapy, occupation, or other responsibility, that, in the opinion of the investigator, would interfere with, or serve as a contraindication to study participation or compliance with the dosing requirements.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2005-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kata L Chillag, PhD, Principal Investigator — Centers for Disease Control and Prevention; Lisa A Grohskopf, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention; Susan Buchbinder, MD, Principal Investigator — San Francisco Dept. of Public Health; Melanie Thompson, MD, Principal Investigator — AIDS Research Consortium of Atlanta; Kenneth H. Mayer, MD, Principal Investigator — Fenway Community Health
Locations (3):
- United States (3):
  - San Francisco Department of Public Health, San Francisco, California
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Fenway Community Health, Boston, Massachusetts

REFERENCES:
- [Derived] Baxi SM, Vittinghoff E, Bacchetti P, Huang Y, Chillag K, Wiegand R, Anderson PL, Grant R, Greenblatt RM, Buchbinder S, Gandhi M, Liu AY. Comparing pharmacologic measures of tenofovir exposure in a U.S. pre-exposure prophylaxis randomized trial. PLoS One. 2018 Jan 9;13(1):e0190118. doi: 10.1371/journal.pone.0190118. eCollection 2018. PMID 29315307
- [Derived] Liu AY, Vittinghoff E, Sellmeyer DE, Irvin R, Mulligan K, Mayer K, Thompson M, Grant R, Pathak S, O'Hara B, Gvetadze R, Chillag K, Grohskopf L, Buchbinder SP. Bone mineral density in HIV-negative men participating in a tenofovir pre-exposure prophylaxis randomized clinical trial in San Francisco. PLoS One. 2011;6(8):e23688. doi: 10.1371/journal.pone.0023688. Epub 2011 Aug 29. PMID 21897852

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in 1/2005 and was completed in 7/2007. Participant follow-up was completed in July 2009.
  Participants were recruited from:
  San Francisco Dept. of Public Health AIDS Research Consortium of Atlanta Fenway Health
Pre-assignment Details: After an initial screening visit, participants were required to meet all enrollment criteria again at the enrollment visit.
Groups:
- Tenofovir Disoproxil Fumarate: Participants received TDF 300mg orally daily for 24 months (immediate arm) or 15 months (delayed arm).
- Placebo: Participants received matching placebo, to be taken daily.
Period: Overall Study
Arm/Group | Tenofovir Disoproxil Fumarate | Placebo
Started | 201 (201 randomized to active drug; 101 to start immediately and 100 after a 9 month delay.) | 199 (199 randomized to placebo; 99 to start immediately and 100 after a 9 month delay.)
Completed | 171 | 160
Not Completed | 30 | 39

BASELINE CHARACTERISTICS:
Population: 400 participants enrolled (200 in San Francisco, 121 in Atlanta, and 79 in Boston). 201 were randomized to TDF and 199 to placebo. Participants were distributed similarly in terms of age, ethnicity, education, no. male partners in previous 3 mo., and no. of unprotected anal sexual contacts within the previous 3 mo.
Groups:
- Tenofovir Disoproxil Fumarate: Active arm: assigned to take TDF, 300mg po daily.
- Placebo: Placebo arm--received matching placebo
- Total: Total of all reporting groups
Arm/Group | Tenofovir Disoproxil Fumarate | Placebo | Total
Number analyzed (Participants) | 201 | 199 | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 201 | 199 | 400
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (9.3) | 36.7 (11.0) | 37.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 201 | 199 | 400
Region of Enrollment [Number; unit: participants]
  United States | 201 | 199 | 400

OUTCOME MEASURES:

1. Primary Outcome: Clinical Safety--Creatinine Elevations
Description: Grade 3 or 4 Creatinine elevations (per National Institutes of Health Division of AIDS toxicity scale)
Time Frame: 24 months (immediate arm) and 15 months (delayed arm)
Population: For biomedical outcomes, a treatment emergent cohort was defined. Participants entered the TE cohort with first dispense and exited with the first occurrence of: (1) completion of follow-up, (2) 30 days after permanent drug interruption, or (3) 30 days after last visit. For delayed arm participants,time before initiation of drug was excluded.
Measure: Number; unit: Participants
Groups:
- Tenofovir Disoproxil Fumarate: TDF, 300 mg orally daily
- Placebo: Matching placebo daily
Arm/Group | Tenofovir Disoproxil Fumarate | Placebo
Number analyzed (Participants) | 186 | 187
Participants | 0 | 0

2. Secondary Outcome: Number of Breakthrough HIV Infections
Description: Number of participants with HIV seroconversions occuring while on study drug
Time Frame: 24 months (immediate arm) and 15 months (delayed arm)
Population: For biomedical outcomes, a treatment emergent cohort was defined which included only those participants who received study drug.
Measure: Number; unit: participants
Arm/Group | Tenofovir Disoproxil Fumarate | Placebo
Number analyzed (Participants) | 186 | 187
participants | 0 | 4

3. Secondary Outcome: Adherence to Study Drug
Description: Estimated exposure to study drug (active and placebo) as assessed by Medication Event Monitoring System (MEMS) caps.
Time Frame: 24 months (immediate arm) and 15 months (delayed arm)
Measure: Number; unit: percentage of doses
Groups:
- Treatment Emergent Cohort: Includes all who entered treatment emergent cohort (active and placebo arms)
Arm/Group | Treatment Emergent Cohort
Number analyzed (Participants) | 373
percentage of doses | 77

4. Secondary Outcome: Behavioral Safety--Unprotected Anal Sex (UAS)
Description: Change in percent of participants reporting unprotected anal intercourse--baseline vs. months 3 through 9 on study.
Time Frame: Nine months
Measure: Number; unit: percentage of ppts reporting UAS
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 400
percentage of ppts reporting UAS | -9

5. Primary Outcome: Clinical Safety--Hypophosphatemia
Description: Grade 3 or 4 hypophosphatemia (per National Institutes of Health Division of AIDS toxicity scale)
Time Frame: 24 months (immediate arm), 15 months (delayed arm)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Tenofovir Disoproxil Fumarate | Placebo
Number analyzed (Participants) | 186 | 187
participants | 1 | 5

6. Other Pre Specified Outcome: >5% Bone Mineral Density Decline at Femoral Neck
Description: Percent of San Francisco participants in the TDF vs. placebo groups who were found to have >5% decline in Bone Mineral Density at the femoral neck.
Time Frame: 24 months (immediate arm), 15 months (delayed arm)
Population: For biomedical outcomes, a treatment emergent cohort was defined which included only those participants who received study drug. In addition, this analysis population includes only those participants for whom bone density analyses were performed.
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir Disoproxil Fumarate | Placebo
Number analyzed (Participants) | 94 | 90
percentage of participants | 13 | 6

ADVERSE EVENTS:
Time Frame: Maximum time period on drug of 24 months for immediate arm participants and 15 months for delayed arm participants.
Description: Treatment emergent cohort: participants enter cohort when study drug is initiated, and exit at the first occurence of one of these events: 1) completion of study visits, 2)30 days after loss to follow up, or 3)30 days after start of permanent drug interruption.
Arm/Group | Tenofovir Disoproxil Fumarate | Placebo
Serious Adverse Events (participants affected / at risk) | 10/186 | 8/187
Other Adverse Events (participants affected / at risk) | 149/186 | 146/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenofovir Disoproxil Fumarate (N=186) | Placebo (N=187)
Depression (Psychiatric disorders) | 1 (4) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenofovir Disoproxil Fumarate (N=186) | Placebo (N=187)
Upper respiratory tract infection (Infections and infestations) | 70 (123) | 67 (127)
Diarrhea (Gastrointestinal disorders) | 33 (42) | 45 (57)
Headache (Nervous system disorders) | 24 (27) | 28 (33)
Depression (Psychiatric disorders) | 17 (21) | 24 (30)
Gastroenteritis (Injury, poisoning and procedural complications) | 19 (24) | 17 (25)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (31) | 12 (14)
Flatulence (Gastrointestinal disorders) | 18 (21) | 18 (22)
Fatigue (General disorders) | 17 (24) | 15 (17)
Nausea (Gastrointestinal disorders) | 20 (27) | 12 (13)
Influenza (Infections and infestations) | 16 (22) | 13 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (21) | 11 (14)
Hypertension (Vascular disorders) | 12 (19) | 9 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 10 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (11) | 13 (16)
Insomnia (Psychiatric disorders) | 10 (10) | 12 (14)
Anxiety (Psychiatric disorders) | 7 (8) | 15 (16)
Dizziness (Nervous system disorders) | 14 (17) | 7 (9)
Herpes simplex (Infections and infestations) | 3 (7) | 12 (15)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 10 (10)
Nasopharyngitis (Infections and infestations) | 6 (8) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All presentations and publications of data from CDC funded studies are subject to CDC clearance prior to publication or presentation.